CLINICAL TRIAL: NCT01900327
Title: Sequential Neoadjuvant Chemoradiotherapy (CRT) Followed by Curative Surgery vs. Primary Surgery Alone for Resectable, Non-metastasized Pancreatic Adenocarcinoma
Brief Title: Neoadjuvant Treatment in Resectable Pancreatic Cancer
Acronym: NEOPA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment failure
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: University Hospital Schleswig-Holstein (Other); Hannover Medical School (Other); St. Josef Hospital Bochum (Other); University of Jena (Other); SRH Wald-Klinikum Gera GmbH (Other); Klinikum Darmstadt (Other); Universität des Saarlandes (Other); Heidelberg University (Other); Staedtisches Klinikum Karlsruhe (Other); University Hospital Freiburg (Other); University Hospital Regensburg (Other); Technical University of Munich (Other); University Hospital Augsburg (Other); Klinikum Stuttgart (Other); Ludwig-Maximilians - University of Munich (Other); University of Rostock (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEOPA
Record Dates: First submitted 2013-06-27; First posted 2013-07-16 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; surgery; chemoradiation; neoadjuvant treatment; overall survival
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Surgical Procedures, Operative; Transurethral Resection of Bladder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- neoadj. Treatment (Experimental): Neoadjuvant CRT with weekly Gemcitabine neoadjuvant 300mg/m2 for 6 weeks combined with external beam radiation (EBRT) delivering a total dose of 50.4 Gy over 28 days in 1.8 Gy fractions will be followed by classical or pylorus-preserving partial pancreato-duodenectomy (PD) and adjuvant chemotherapy (CTx), preferentially using Gemcitabine adjuvant (1000 mg/m2 6 cycles at day 1, 8, 15 of each 28-day cycle).
  Interventions: Radiation: External Beam Radiation; Drug: Gemcitabine neoadjuvant; Procedure: Surgery; Drug: Gemcitabine adjuvant
- Upfront Surgery (Active Comparator): Upfront PD followed by adjuvant CTx, preferentially with Gemcitabine adjuvant (1000 mg/m2 6 cycles at day 1, 8, 15 of each 28-day cycle).
  Interventions: Procedure: Surgery; Drug: Gemcitabine adjuvant

INTERVENTIONS:
Radiation: External Beam Radiation — Neoadjuvant CRT with external beam radiation (EBRT) delivering a total dose of 50.4 Gy over 28 days in 1.8 Gy fractions.
  Other Names: External Beam Radiation Therapy; EBRT
  Arms: neoadj. Treatment
Drug: Gemcitabine neoadjuvant — weekly Gemcitabine 300mg/m2 for 6 weeks neoadjuvant
  Other Names: Gemcitabin; Gemzar
  Arms: neoadj. Treatment
Procedure: Surgery — Upfront pancreato-duodenectomy
  Other Names: Tumor resection
Drug: Gemcitabine adjuvant — Postoperative adjuvant Chemotherapy preferentially using Gemcitabine (1000 mg/m2 6 cycles at day 1, 8, 15 of each 28-day cycle. Administered in both arms, experimental AND active comparator
  Other Names: Gemcitabin; Gemzar; 2',2'-Difluordesoxycytidin

SUMMARY:
Sequential Neoadjuvant Chemoradiotherapy (CRT) Followed by Curative Surgery vs. Primary Surgery Alone for Resectable, Non-metastasized Pancreatic Adenocarcinoma

DETAILED DESCRIPTION:
Median overall-survival (OS) after surgery in curative intent for non-metastasized pancreas cancer ranges under study conditions from 17.9 months to 23.6 months. Tumor recurrence occurs locally, at distant sites (liver, peritoneum, lungs), or both. Observational and autopsy series report local recurrence rates of up to 87% even after potentially "curative" R0 resection. To achieve better local control, neoadjuvant chemo-radiation therapy (CRT) has been suggested for preoperative tumour downsizing, to elevate the likelihood of curative, margin-negative R0 resection and to increase the OS rate. However, controlled, randomized trials addressing the impact of neoadjuvant CRT survival do not exist. The underlying hypothesis of this randomized, two-armed, open-label, multicenter, phase III trial is that neoadjuvant CRT increases the three-year overall survival by 12% (30% to 42%) compared to patients undergoing upfront surgery for resectable pancreatic cancer. Overall, 410 patients (n=205 in each study arm) will be enrolled in the trial, taking into regard an expected drop out rate of 7% and allocated either to receive neoadjuvant CRT prior to surgery or to undergo surgery alone. Circumferential resection margin status, i.e. R0 and R1 rates, respectively, surgical resectability rate, local and distant disease-free and global survival, and first site of tumor recurrence constitute further essential endpoints of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Histology-proven adenocarcinoma of the pancreatic head/uncinate process with a tumor size greater 2 cm (≥cT2) and/or close contact to the superior mesenteric vessels (≤3 mm in preoperative staging).
* No evidence of metastasis to distant organs (liver, peritoneum, lung, others).
* For determination of resectability, a multi-detector CT (MDCT) with at least 16 rows applying both oral and intravenous contrast media is performed. MDCT-based imaging focuses on the upper abdomen with native, arterial, and parenchyma phase, where the parenchyma phase should include the pelvis. Imaging criteria derived from the recent consensus definition of the Society of Surgical Oncology, the American Society of Clinical Oncology and the American Hepato-Pancreatico-Biliary Association [1] are applied for preoperative assessment of local resectability.
* Potential Resectability: visualizable fat plane around celiac and superior mesenteric arteries, and patent superior mesenteric/portal vein (SMV/PV).
* Borderline Resectability: substantial superior mesenteric/portal vein impingement, tumor abutment on the SMA < 180°, GDA encasement up to the origin of the hepatic artery, or colonic/mesenteric root invasion.
* Karnofsky performance status ≥ 80%
* Serum creatinine level ≤ 3.0 mg/dl
* Serum total bilirubin level ≤ 3.0 mg/dl in the absence of biliary obstruction (In the event of biliary obstruction, patients allocated to the CRT group must undergo interventional endoscopy or percutaneous drainage for biliary decompression. Post-interventionally, bilirubin levels should be ≤ 3.0 mg/dl before patients are subjected to CRT. In control patients undergoing upfront surgery, serum total bilirubin levels ≤ 10.0 mg/dl are tolerated, unless clinical and laboratory signs of severe cholangitis take place. Patients with serum total bilirubin level > 10.0 mg/dl undergo preoperative biliary decompression, preferentially by interventional endoscopy)
* White blood cell count ≥ 3.5 x 109/ml, platelet count ≥ 100 x 109/ml
* Ability to understand and willingness to consent to formal requirements for study participation
* Written informed consent

Exclusion Criteria:

* Age ≤ 18 years
* Neuroendocrine, acinar cancer
* Cancers of the pancreatic body or tail, i.e. lesions left to the SMV
* Recurrent disease
* Infiltration of extrapancreatic organs (except duodenum and transverse colon)
* Persistent cholestasis/cholangitis despite adequate biliary stenting
* Gastric outlet obstruction, especially in the event of endoscopically evidenced tumor invasion into the gastroduodenal mucosa.
* Tumor specific pre-treatment
* History of gastrointestinal perforation, e.g. perforated colonic diverticulitis, abdominal abscess or intestinal fistula within 6 months prior to potential study participation
* Radiographic evidence of severe portal hypertension/cavernomatous transformation that may, at the discretion of the participating investigators, hamper surgery
* Other concurrent malignancies except for basal cell cancer of the skin and in-situ cervical cancer
* Premalignant hematologic disorders, e.g. myelodysplastic syndrome
* Severe organ dysfunctions (e.g. Liver cirrhosis ≥ Child B; Cardio-pulmonal diseases (NYHA ≥III, arrhythmia Lown III/IV, global respiratory insufficiency); Ascites; Acute pancreatitis; bleeding diathesis, coagulopathy, need for full-dose anticoagulation or INR > 1.5; other severe diseases that might prevent completion of the treatment regimen)
* Chronic infectious diseases, especially immune deficiency syndromes, e.g. HIV infection, active tuberculosis within 12 months prior to potential study participation
* History of severe neurologic disorders, e.g. cerebrovascular ischemia
* History of prior deep venous thrombosis or pulmonary embolism
* Pregnant or nursing women are ineligible and patients of reproductive potential must agree to use an effective contraceptive method during participation in this trial and for 6 months following the trial
* Serious medical, psychological, familial, sociological or geographical conditions or circumstances potentially hampering compliance with the study protocol and follow-up Participation in other clinical trials during the last 6 months before allocation to trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-02; Primary Completion 2016-11-22 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
3-Year Survival Rate | 3 years after last patient in
  Primary outcome measure is the efficacy of neoadjuvant CRT in improving 3-year survival probability from 30% in the control arm undergoing upfront surgery without neoadjuvant CRT to 42% (relative increase of 40%) in the study arm undergoing CRT. The underlying guess of a 30% 3-year survival probability in the control group derives from an assumed median overall survival (MOS) of 20.7 months which corresponds with a MOS of 17.9 months to 23.6 months reported in several randomized trials.

SECONDARY OUTCOMES:
R0 Resection rate | 3 days
  Histology-proven R0 resection rate based on a standardized histopathological handling of the surgical specimen.
Frequency of Toxicity Events | three years
  Frequency of moderate and severe toxicity events and drop-out rate due to therapy related toxicity (NCI Common Toxicity Criteria v2.0)
Resectability rate | one day
  Resectability rate
Rate of intraoperative irregularities | one day
  Rate of unexpected intraoperative irregularities, operative time, blood transfusion requirement, postoperative morbidity rate, especially that of pancreatic fistula, and mortality rate
Postoperative Complications | three months
  Rate of patients with severe postoperative complications (postoperative recovery > 8 weeks) rendering adjuvant treatment worthless
Disease progression during neoadjuvant therapy | three months
  Rate of patients with disease progression during neoadjuvant therapy (only applicable in treatment arm)
Quality of life | three years
  Quality of life analysis (EORTC QLQ C30 questionnaire). Assessment of QLQ after completion of neoadjuvant RCTx, after surgery (before hospital discharge) and 6, 12 and 18 months after completion of treatment
Disease-free Survival | three years
  Median disease-free survival (DFS, local and distant), overall survival (OS)
First site of tumor recurrence | two years
  First site of tumor recurrence as determined by abdominal computed tomography during follow-up study visits

CONTACTS AND LOCATIONS:
Overall Officials: Jakob R Izbicki, MD, FACS, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (16):
- Germany (16):
  - University Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Heidelberg University, Heidelberg, Baden-Wurttemberg
  - Technische Universität München, München, Bavaria
  - University Regensburg, Regensburg, Bavaria
  - Klinikum Augsburg, Augsburg, Bayer
  - Klinikum Darmstadt, Darmstadt, Hesse
  - Hannover Medical School, Hanover, Lower Saxony
  - University of Rostock, Rostock, Mecklenburg-Vorpommern
  - St. Joseph Hospital Bochum, Bochum, North Rhine-Westphalia
  - Saarland University, Homburg, Saarland
  - University of Schleswig-Holstein Kiel, Kiel, Schleswig-Holstein
  - University of Schleswig-Holstein Lübeck, Lübeck, Schleswig-Holstein
  - Klinikum Gera, Gera, Thuringia
  - University of Jena, Jena, Thuringia
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Klinikum Karlsruhe, Karlsruhe

REFERENCES:
- [Derived] Tachezy M, Gebauer F, Petersen C, Arnold D, Trepel M, Wegscheider K, Schafhausen P, Bockhorn M, Izbicki JR, Yekebas E. Sequential neoadjuvant chemoradiotherapy (CRT) followed by curative surgery vs. primary surgery alone for resectable, non-metastasized pancreatic adenocarcinoma: NEOPA- a randomized multicenter phase III study (NCT01900327, DRKS00003893, ISRCTN82191749). BMC Cancer. 2014 Jun 7;14:411. doi: 10.1186/1471-2407-14-411. PMID 24906700
- See also: Homepage University Medical Center — http://www.uke.de